CLINICAL TRIAL: NCT06521099
Title: A Novel Conditioning Approach to Counter Loneliness in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG Man Lok Nichol, Assistant Professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2022-2023-0082
Record Dates: First submitted 2024-07-11; First posted 2024-07-25 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Loneliness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluative conditioning group with positive stimuli (Experimental): Participants will be exposed to social stimuli paired with positive stimuli across multiple sessions.
  Interventions: Behavioral: Evaluative Conditioning with positive stimuli
- Control group with neutral stimuli (Active Comparator): Participants will be exposed to social stimuli paired with neutral stimuli across multiple sessions.
  Interventions: Behavioral: Conditioning with neutral stimuli

INTERVENTIONS:
Behavioral: Evaluative Conditioning with positive stimuli — In the pre-conditioning phase, participants will be exposed to pictures that vary in their emotional (negative, positive) and social (non-social, social) content. For each picture, they are required to indicate their immediate perceived valence (between negative to positive), degree of social motivation (between none to high) on Likert-scales. In the conditioning phase, emotional social pictures will be selected and paired with non-social positive stimuli for trials in random order, for 6 sessions across 3 weeks. In the post-conditioning phase, participants will be asked to evaluate the valence of the stimuli again similar to that in pre-conditioning phase.
  Arms: Evaluative conditioning group with positive stimuli
Behavioral: Conditioning with neutral stimuli — In the pre-conditioning phase, participants will be exposed to pictures that vary in their emotional (negative, positive) and social (non-social, social) content. For each picture, they are required to indicate their immediate perceived valence (between negative to positive), degree of social motivation (between none to high) on Likert-scales. In the conditioning phase, emotional social pictures will be selected and paired with with neutral non-social stimuli for trials in random order, for 6 sessions across 3 weeks. In the post-conditioning phase, participants will be asked to evaluate the valence of the stimuli again similar to that in pre-conditioning phase.
  Arms: Control group with neutral stimuli

SUMMARY:
This study aims to test the efficacy of a 6-session conditioning paradigm by investigating the conditioning-induced change in the socio-affective processing, loneliness, depressive symptoms, and neural correlates of lonely adults.

DETAILED DESCRIPTION:
Potential participants will first be invited to complete a loneliness questionnaire online. Lonely adults will then be invited to undergo further screening. At baseline prior to the intervention training sessions, participants will first complete tests and questionnaires on loneliness, mood and depressive symptoms in addition to other socio-affective measures, and they will also be invited to receive resting-state functional MRI scanning in a 3T MRI scanner. Participants will then be allocated to one of the two intervention arms (the evaluative conditioning, and the control) in a randomized fashion with approximately half in each group. They will then complete the pre-conditioning phase of the allocated intervention arm, and their ratings on the stimuli presented during this phase will be assessed. In the conditioning phase, they will be invited to attend 6 sessions. After completing the conditioning phase, participants will be invited to complete the post- conditioning phase, providing ratings on the stimuli like the pre-conditioning phase. Immediately after, and also 3 months after, participants will be invited to complete again tests and questionnaires on loneliness, mood and depressive symptoms in addition to other socio-affective measures, and they will also be invited to receive resting-state functional MRI scanning in a 3T MRI scanner.

ELIGIBILITY:
Inclusion Criteria:

* No histories of learning impairment, major psychiatric disorders or neurological disorders other than depression
* Normal intelligence
* At least primary school education

Exclusion Criteria:

* On medication or treatments within 2 weeks prior to the beginning of the study that would affect the individual's brain, cognitive and affective functions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Self-reported loneliness | Baseline, immediately after, and 3 months after the intervention
  Loneliness is assessed based on the UCLA loneliness scale (Version 3), a 20-item 4-point Likert scale (score range 20 - 80) in which higher scores indicate greater degrees of loneliness.
Implicit loneliness | Baseline, immediately after, and 3 months after the intervention
  Implicit loneliness will be measured by Implicit Association Test about the relative strength of association between our participants' target concept 'Self' and attribute 'Lonely'.

SECONDARY OUTCOMES:
Valence of social stimuli | Baseline, immediately after, and 3 months after the intervention
  For each stimuli, they are required to indicate their immediate perceived valence (between negative to positive) of the scenes on a 7-point Likert scale (1 = strongly positive, 7 = strongly negative).
Social motivation towards social stimuli | Baseline, immediately after, and 3 months after the intervention
  For each stimuli, they are required to indicate their immediate perceived degree of social motivation (between none to high) of the scenes on a 7-point Likert scales (1 = no, 7 = very high).
Loneliness-related activation patterns and connectivity in neural networks | Baseline, immediately after, and 3 months after the intervention
  Neural connectivity in Default Mode Network, Ventral Attention Network, Frontoparietal Network are assessed by fMRI
Depressive symptoms | Baseline, immediately after, and 3 months after the intervention
  Depressive symptoms are assessed based on the Hospital Anxiety and Depression Scale, a 14-item scale assessing severity of depressive and anxiety symptom (score range 0 - 21 for both subscale), with higher scores indicating higher severity
Daily loneliness | Through study completion, on average of 4 months
  Daily loneliness is assessed based on a 5-minute self-report on a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Nichol ML Wong, PhD, Principal Investigator — Education University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong NML, Lee TMC. Evaluating the effects of a conditioning training paradigm on loneliness, socio-affective processing, and brain connectivity: a study protocol of a two-arm randomised controlled trial. BMC Psychol. 2025 Aug 27;13(1):975. doi: 10.1186/s40359-025-03342-3. PMID 40866945